CLINICAL TRIAL: NCT05307653
Title: The Analgesic Effect Of Sacral Erector Spinae, Penile And Caudal Block For Pain Relief After Hypospadius Surgery: Randomized Controlled Study
Brief Title: Sacral Erector Spinae,Penile and Caudal Block for Pain Relief After Hypospadias Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Amr Arafa Elbadry, Principle Investigator, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pain Relief After Hypospadius
Record Dates: First submitted 2022-03-23; First posted 2022-04-01 (Actual); Last update posted 2022-09-02 (Actual); Status verified 2022-08

CONDITIONS: Sacral Erector Spinae, Penile And Caudal Block For Pain Relief After Hypospadius Surgery

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Penile block (Experimental): Penile block was performed in supine position. The penis was retracted caudally and then fixed with a leucoplast. After identifying the symphysis pubis (SP), a 22-gauge needle was inserted vertically about 1 cm lateral to the SP, and bupivacaine 0.5% (0.1 ml/kg, maximum 2.5 ml) was injected on each side after penetrating the Scarpa's fascia.
  Interventions: Procedure: Penile block
- Erector spinea plain block group (Experimental): Ultrasound guided ESPB was performed in prone position by Philips © (CX50 Extreme edition). The superficial probe was placed longitudinally at the midline just above the sacrum, and both erector spinae muscles and median sacral crests were identified. Using the in-plane approach, a 22-gauge needle was inserted in a craniocaudal direction till reaching the tip of the fourth median sacral crest. After negative aspiration to avoid intravascular or intrathecal puncture, bupivacaine 0.25% (1 ml/kg, maximum 20 ml) was administered.
  Interventions: Procedure: Erector spinea plain block
- Caudal group (Experimental): Caudal block was performed in the left lateral position. A 22 G needle was inserted through the sacral hiatus. The loss of resistance method was used to pass through the sacrococcygeal membrane and enter the caudal epidural space. Negative aspiration was then performed. When no blood or cerebrospinal fluid was observed, bupivacaine 0.25% (1 ml/kg, maximum 20 ml) was administered. The patient was returned to the supine position after the procedure was completed.
  Interventions: Procedure: Caudal block

INTERVENTIONS:
Procedure: Penile block — Penile block was performed in supine position. The penis was retracted caudally and then fixed with a leucoplast. After identifying the symphysis pubis (SP), a 22-gauge needle was inserted vertically about 1 cm lateral to the SP, and bupivacaine 0.5% (0.1 ml/kg, maximum 2.5 ml) was injected on each side after penetrating the Scarpa's fascia.
  Arms: Penile block
Procedure: Erector spinea plain block — Ultrasound guided ESPB was performed in prone position by Philips © (CX50 Extreme edition). The superficial probe was placed longitudinally at the midline just above the sacrum, and both erector spinae muscles and median sacral crests were identified. Using the in-plane approach, a 22-gauge needle was inserted in a craniocaudal direction till reaching the tip of the fourth median sacral crest. After negative aspiration to avoid intravascular or intrathecal puncture, bupivacaine 0.25% (1 ml/kg, maximum 20 ml) was administered.
  Arms: Erector spinea plain block group
Procedure: Caudal block — Caudal block was performed in the left lateral position. A 22 G needle was inserted through the sacral hiatus. The loss of resistance method was used to pass through the sacrococcygeal membrane and enter the caudal epidural space. Negative aspiration was then performed. When no blood or cerebrospinal fluid was observed, bupivacaine 0.25% (1 ml/kg, maximum 20 ml) was administered. The patient was returned to the supine position after the procedure was completed.
  Arms: Caudal group

SUMMARY:
Caudal anaesthesia is recommended for most surgical procedures of the lower part of the body, mainly below the umbilicus, including inguinal hernia repair, urinary and digestive tract surgery and orthopaedic procedures on the pelvic girdle and lower extremities.

It has been well established that a dorsal penile nerve block immediately after surgery decreases postoperative pain in children undergoing hypospadias repair. For decades, penile block was widely and effectively used for various types of penile reconstructive surgery.

Recently, due to improved composition, dosage and concentration of local anaesthetics and low incidence of negative side effects, such as motor blockade and postoperative nausea and vomiting, caudal anaesthesia has become one of the most used and accepted regional blocks for children undergoing hypospadias repair.

However, postoperative patient comfort is a major issue after distal hypospadias repair and depends on adequate analgesia and unimpaired micturition, especially when no suprapubic catheter is in place. Micturition impairment and urinary retention is a known side effect of caudal block anaesthesia.

The comparison of penile block and caudal block has not been described in the literature to our knowledge.

Use of ESPB for different indications from different levels has become the new trend of regional anesthesia practice from the moment it was first defined . There have been many reports for its use in thoracic and lumbar levels.

This great interest probably depends on its effectiveness as well as the ease of the block technique: injecting the local anesthetic deep to the erector spinae muscle (ESM) above the transverse process. With this report, we would like to identify a modification to sacral ESPB with our longitudinal midline approach with the presentation of a case of an infant who was scheduled for hypospadias repair.

DETAILED DESCRIPTION:
Patients will be randomly divided into three groups by using a computer-generated randomization. Sealed opaque envelopes containing group allocation will be before the blocks will be performed. Then, each patient will be asked to choose one of the envelopes and give to an anesthesiologist who will compare it to the computer-generated list and hence assignee her to one of the three groups. Anesthesiologist (who will be blinded to the collected data until the end of the study) will perform the block techniques and administer the medication.

* Group C (Caudal group) n=44: after prep and drep, in left lateral position caudal block will be performed with bupivacaine 0.25%, 1 ml/kg (max 20 ml).
* Group P (Penile block) n=44: after prep and drep in supine position, the penis will be retracted downward and fixed with leucoplast. The markers for injection will be, symphysis pubis, 0.5 to 1 cm lateral to the midline, the needle will be inserted vertically (medially-caudally) until penetrating fascia scarpa and bupivacaine 0.5%, 0.1 ml/kg (max 2.5 ml), will be injected in each side. Blocks will be performed with 22-G needles and skin incision will be performed 20 minutes after block in each group.
* Group E (Erector spinea plain block group) n=44:

Before the start of surgery, patient will be turned to prone position for block application. Following cleansing of the block area, linear ultrasound probe (Esaote My Lab 6 US machine, Florence, Italy) will be placed longitudinally to midline just above the sacrum . Median sacral crests and erector spinae muscle will be identified.

A 22G, 50mm needle (B. Braun Melsungen, Germany) will be inserted from the edge of the probe using in-plane technique. Needle will be advanced with a cranial to caudal direction until its tip touched to the top of the 4th median sacral crest. Following negative aspiration, 8 mL of 0, 25% Bupivacaine (with a dose of 1 mL/kg) will be injected for the block application. Then the patient will be turned to supine position and surgery started.

Anesthesia Protocol All the patients will be adequately assessed preoperatively in the anesthesia clinic through history taking, general and local examination, and requesting investigation. Adequate explanation of the procedure, benefit, and potential hazards will be done to the parents with final reassurance of them. All children will receive sedation in the form of oral midazolam 0.05 mg/kg 15 minutes before admission to the operating room.

Upon admission to the operating room, intravascular access will be obtained with starting i.v infusion of Dextrose 5% in normal saline (7 ml/kg). Then, the patients will be attached to a monitor of pulse oximetry, non-invasive blood pressure, end-tidal carbon dioxide, temperature, and 5 leads electrocardiogram. Induction of anesthesia will be carried out using sevoflurane 6% in oxygen: air (4:1) till the child loss the consciousness, then, fentanyl 0.5 ug/kg will be given intravenously and atracurium 1 ug/kg will be given intravenously to facilitate endotracheal intubation. A suitable sized endotracheal tube will be introduced and secured with connection of the patients to a mechanical ventilator (pressure-controlled mode) which parameters will be adjusted to maintain end-tidal carbon dioxide 36-40 mmHg.

Anesthesia will be maintained by sevoflurane (1 MAC) with incremental doses of atracurium. Also, incremental doses of fentanyl 0.5 ug/kg will be given i.v in case of increase bispectral index (BIS) more than 60 or by increase in the heart rate or the mean arterial pressure by more than 20% of the baseline values.

At the end of the surgery, the sevoflurane will be switched off with reversal of the muscle relaxation by combination of neostigmine 0.04 mg/kg and atropine 0.01 mg/kg. Awake extubation will be then performed with transporting the child to the recovery room for adequate postoperative monitoring. All the children will receive paracetamol 15 mg/kg i.v infusion every 6 h. The children will be discharged from the recovery room when their modified Aldrete's score reach 10.

Postoperatively, patient was evaluated with Face, Leg, Activity, Cry, Consolability Revised (FLACC-R) score for pain management and it was 0 or 1 for entire postoperative 24 h. In recovery or ward, rectal acetaminophen was administered for an age-appropriate pain score between 3 and 5 (0-10) and intravenous meperidine 1 mg/kg for an age-appropriate pain score of >5 (0-10).

Measurements The following parameters will be recorded by an anesthesia resident not included in the study and blinded to its groups: -

* Demographic data (Age in month, body weight, and ASA class)
* Total consumption of pethidine (mg/kg) in first day postoperatively. (secondary outcome)
* The duration of postoperative analgesia which defied as: The time (in hours)from the beginning of the block to the first rescue analgesia request (primary outcome)
* The postoperative pain score (FLAC pain score) every 2 hours in the first 8 hours then every 4 hours till 24 h. (Secondary outcome)
* The total dose of fentanyl consumed intraoperatively.
* The incidence of perioperative complications including bradycardia, hypotension, nausea and vomiting, localized hematoma, infection, or pruritis.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria was patients with distal penile, subcoronal and coronal type of hypospadias, scheduled for repair with an intermittent non-dribbling urethral stent for 7 days or less.

Exclusion Criteria:

* Bleeding diathesis
* Known allergy to local anesthesia medications
* Active infection at the injection area
* History of developmental delay
* Mental retardation (due to difficult pain assessment).

Ages: 1 Year to 5 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes
Enrollment: 132 (Actual)
Dates: Start 2022-04-15 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2022-08-30 (Actual)

PRIMARY OUTCOMES:
Time to the first analgesic request | 24 hours postoperative
  The time (in hours) from the beginning of the block to the first rescue analgesia request was recorded

SECONDARY OUTCOMES:
Face, Legs, Activity, Cry, and Consolability (FLACC) Score | 24 hours Postoperative
  FLACC scale will be used to assess pain for children between the ages 2 months and 7 years or individuals that unable to communicate their pain. The scale is scored of 0-10 with 0 representing no pain. The scale has five criteria, which are each assigned a score of 0, 1or 2. FLACC scale will be recorded every 2 hours in the first 8 hours then every 4 hours till 24 h. (Secondary outcome)
The total amount of analgesia | 24 hours Postoperative
  Total consumption of pethidine (mg/kg) in the first day postoperatively
The incidence of perioperative complications. | 24 hour postoperatively
  The incidence of perioperative complications including bradycardia, hypotension, nausea and vomiting, localized hematoma, infection, or pruritis was recorded.
Penile engorgement | Intraoperatively
  The occurence of penile engorgement.

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University Hospitals, Tanta, ELgharbiaa, Egypt